CLINICAL TRIAL: NCT05723172
Title: 40Hz tACS in Treating Cognitive Function and Modulating Neurophysiology of Patients With Alzheimer's Disease: a Triple Blind Randomized Sham-controlled Trial
Brief Title: 40Hz tACS in Treating Cognitive Function and Modulating Neurophysiology of Patients With Alzheimer's Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Che-Sheng Chu (Other)
Responsible Party: Sponsor-Investigator, Che-Sheng Chu, Attending Physician, Kaohsiung Veterans General Hospital.
Organization: Kaohsiung Veterans General Hospital. (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: VGHKS-112-01
Record Dates: First submitted 2023-01-25; First posted 2023-02-10 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Alzheimer Disease
Keywords: Alzheimer's disease; tACS
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- active tACS (Active Comparator): 40 mins tACS for 10 consecutive daily sessions
  Interventions: Device: active tACS
- sham tACS (Sham Comparator): 40 mins sham tACS for 10 consecutive daily sessions
  Interventions: Device: sham tACS

INTERVENTIONS:
Device: active tACS — 40 mins tACS for 10 consecutive daily sessions
  Arms: active tACS
Device: sham tACS — 40 mins sham tACS for 10 consecutive daily sessions
  Arms: sham tACS

SUMMARY:
Gamma brain activity is crucial for cognitive function and intra-brain communication. Gamma frequency stimulation via transcranial alternating current stimulation(tACS) might alleviate memory deficits on both animal models of Alzheimer's disease (AD) and clinical trial. The study aims to assess the safety and efficacy of tACS on cognitive function and modulating neurophysiology in patients with AD.

DETAILED DESCRIPTION:
Gamma brain activity is crucial for cognitive function and intra-brain communication. Gamma frequency stimulation via transcranial alternating current stimulation(tACS) might alleviate memory deficits on both animal models of Alzheimer's disease (AD) and clinical trial. The study aims to assess the safety and efficacy of tACS on cognitive function and modulating neurophysiology in patients with AD.

40mins 10Hz-tACS for daily consecutive sessions will be given.

ELIGIBILITY:
Inclusion Criteria:

* aged 60- to 90-year-old
* clinical dementia rating scale (CDR) of 1 or mini-mental state examination (MMSE) score of 18 to 26.
* Participants were allowed to maintain their anti-dementia medications without changes from at 3 months before and throughout the study.

Exclusion Criteria:

* having contraindications for tACS, e.g., implanted brain medical devices or mental in the head, having arrhythmia and with pacemaker implantation, having history of seizures, having history of intracranial neoplasms or surgery, or severe head injuries or cerebrovascular diseases
* clinical depression measured by Hamilton depression rating scale score equal and over 17

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Alzheimer's Disease Assessment Scale-Cognitive Subscale, ADAS-Cog | Change from baseline, two weeks, and one months follow-up
  The ADAS-Cog consists of items from the following areas chosen for their sensitivity to Alzheimer's disease: language; memory; praxis; and orientation. The test takes 30-35 minutes to administer and the item scores generally range from 1-5.

SECONDARY OUTCOMES:
Wechsler adult intelligence scale, WAIS-IV, digit span | Change from baseline and two weeks
  The Wechsler Adult Intelligence Scale (WAIS) is an IQ test designed to measure intelligence and cognitive ability in adults and older adolescents. It is currently in its fourth edition (WAIS-IV) released in 2008 by Pearson, and is the most widely used IQ test, for both adults and older adolescents, in the world. We used WAIS-IV, digit span subscale, to examine attention among subjects; Digit span was by listening to sequences of numbers orally and to repeat them as heard, in reverse order, and in ascending order.
Wechsler adult intelligence scale, WAIS-IV, digit symbol coding | Change from baseline and two weeks
  We used WAIS-IV, digit symbol coding subscale, to examine processing speed among subjects; The digit symbol coding is a paper-and-pencil cognitive test presented on a single sheet of paper that requires a subject to match symbols to numbers according to a key located on the top of the page. The subject copies the symbol into spaces below a row of numbers. The number of correct symbols within the allowed time, usually 90 to 120 seconds, constitutes the score
Wechsler adult intelligence scale, WAIS-IV, vocabulary | Change from baseline and two weeks
  We used WAIS-IV, vocabulary subscale, to examine language function among subjects; The vocabulary subtest requires the client to try to define up to 30 words. This subtest assesses the client's understanding of words and reflects: language development, expressive language skills, cultural and educational experiences, ability to use words appropriately, retrieval of information from long-term memory.
Subjective Cognitive Decline Questionnaire: SCD-QMyCog | Change from baseline and two weeks
  The SCD-Q is a validated questionnaire that assesses the presence of a subjective cognitive decay in abilities such as memory, attention, language or executive functions. This scale is made up of two parts: MyCog is filled by the subject, TheirCog by the caregiver. Both parts have 24 identical dichotomous questions (yes/no), that evaluate decline for memory performances, language and executive functions in the last 2 years of daily life. The SCD-Q score for MyCog and TheirCog ranges from 0 to 24, with higher scores associated with greater perceived cognitive changes (cut to be classified as SCD = 7).
Neuropsychiatric Inventory (NPI) | Change from baseline and two weeks
  The Neuropsychiatric Inventory (NPI) was developed to assess dementia-related behavioral symptoms. The NPI examined 12 sub-domains of behavioral functioning: delusions, hallucinations, agitation/aggression, dysphoria, anxiety, euphoria, apathy, disinhibition, irritability/lability, aberrant motor activity, night-time behavioral disturbances and appetite and eating abnormalities
Mini-Mental State Examination, MMSE | Change from baseline and two weeks
  A Mini-Mental State Examination (MMSE) is a set of 11 questions that doctors and other healthcare professionals commonly use to check for cognitive impairment (problems with thinking, communication, understanding and memory). The maximum score for the MMSE is 30. A score of 25 or higher is classed as normal. If the score is below 24, the result is usually considered to be abnormal, indicating possible cognitive impairment.
HRV (heart rate variability) | Change from baseline, after one session, and two weeks
  Heart rate variability (HRV) is the physiological phenomenon of variation in the time interval between heartbeats. It is measured by the variation in the beat-to-beat interval. By measuring HRV, it reflects individual's sympathetic and parasympathetic tone.
peripheral amyloid beta and tau related markers | Change from baseline and two weeks
  Peripheral Amyloid beta and tau protein as risk biomarkers of Alzheimer's disease. We check this to see the influence of tACS on AD-related biomarkers
EEG (electroencephalogram) | Change from baseline, after one session, and two weeks
  An electroencephalogram (EEG) is a recording of brain activity. During this painless test, small sensors are attached to the scalp to pick up the electrical signals produced by the brain.
  We will check time and/or frequency domain EEG characteristics between those receiving active and sham intervention at different time follow-up points

CONTACTS AND LOCATIONS:
Overall Officials: Che-Sheng Chu, MD, Principal Investigator — Department of Psychiatry, Kaohsiung Veterans General Hospital, Taiwan
Locations (1):
- Department of Psychiatry, Kaohsiung Veterans General Hospital, Kaohsiung City, Taiwan

REFERENCES:
- [Background] Ching PY, Hsu TW, Chen GW, Pan CC, Chu CS, Chou PH. Efficacy and Tolerability of Cranial Electrotherapy Stimulation in the Treatment of Anxiety: A Systemic Review and Meta-Analysis. Front Psychiatry. 2022 Jun 9;13:899040. doi: 10.3389/fpsyt.2022.899040. eCollection 2022. PMID 35757229
- [Background] Chou PH, Lin YF, Lu MK, Chang HA, Chu CS, Chang WH, Kishimoto T, Sack AT, Su KP. Personalization of Repetitive Transcranial Magnetic Stimulation for the Treatment of Major Depressive Disorder According to the Existing Psychiatric Comorbidity. Clin Psychopharmacol Neurosci. 2021 May 31;19(2):190-205. doi: 10.9758/cpn.2021.19.2.190. PMID 33888649
- [Background] Chu CS, Li CT, Brunoni AR, Yang FC, Tseng PT, Tu YK, Stubbs B, Carvalho AF, Thompson T, Rajji TK, Yeh TC, Tsai CK, Chen TY, Li DJ, Hsu CW, Wu YC, Yu CL, Liang CS. Cognitive effects and acceptability of non-invasive brain stimulation on Alzheimer's disease and mild cognitive impairment: a component network meta-analysis. J Neurol Neurosurg Psychiatry. 2021 Feb;92(2):195-203. doi: 10.1136/jnnp-2020-323870. Epub 2020 Oct 28. PMID 33115936
- [Background] Chen GW, Hsu TW, Ching PY, Pan CC, Chou PH, Chu CS. Efficacy and Tolerability of Repetitive Transcranial Magnetic Stimulation on Suicidal Ideation: A Systemic Review and Meta-Analysis. Front Psychiatry. 2022 May 6;13:884390. doi: 10.3389/fpsyt.2022.884390. eCollection 2022. PMID 35599760
- [Background] Hung YY, Yang LH, Stubbs B, Li DJ, Tseng PT, Yeh TC, Chen TY, Liang CS, Chu CS. Efficacy and tolerability of deep transcranial magnetic stimulation for treatment-resistant depression: A systematic review and meta-analysis. Prog Neuropsychopharmacol Biol Psychiatry. 2020 Apr 20;99:109850. doi: 10.1016/j.pnpbp.2019.109850. Epub 2019 Dec 19. PMID 31863873